CLINICAL TRIAL: NCT01389193
Title: Targeting Glial Inhibition to Attenuate Chronic Migraine: AN INTERNATIONAL DOUBLE-BLIND, RANDOMISED, PLACEBO-CONTROLLED TRIAL OF IBUDILAST
Brief Title: Ibudilast in the Treatment of Patients With Chronic Migraine.
Acronym: IBU-003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parisa Gazerani (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Migraine Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Parisa Gazerani, Associtae professor, Aalborg University
Organization: Aalborg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IBU-003; MRF and DRC (Other Grant/Funding Number: Migraine Research Foundation, Danish Research Council)
Record Dates: First submitted 2011-06-29; First posted 2011-07-08 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Migraine Headache
Keywords: ibudilast; migraine; glial cell
MeSH Terms: conditions — Migraine Disorders | interventions — ibudilast; Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibudilast (Experimental)
  Interventions: Drug: Ibudilast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibudilast — Ibudilast 40 mg twice daily oral capsules for a duration of 8 weeks
  Other Names: Ibudilast (Ketas® 10 mg capsules) manufactured by Kyorin Pharmaceuticals.
  Arms: Ibudilast
Drug: Placebo — Placebo 40 mg twice daily oral capsules for a duration of 8 weeks
  Other Names: Pharmaceutical Packaging Professionals, West Thebarton Rd, Thebarton, South Australia
  Arms: Placebo

SUMMARY:
This will be a double-blind, randomised, placebo-controlled, two period cross over study of ibudilast in the treatment of chronic migraine.

For participants resident in Adelaide, South Australia (i.e. "local participants"):

The study will involve a screening visit followed by eight visits to the Pain and Anaesthesia Research Clinic (PARC), within the Royal Adelaide Hospital (RAH), for baseline testing, initiation of the study medications and ongoing data collection (one baseline and three study visits during each treatment period).

At the baseline visit, blood samples to assess biomarkers (glutamate, calcitonin gene-related peptide, glial fibrillary acidic protein and S100β) will be taken. Patients will then be randomised (in a 1:1 ratio) to commence either ibudilast or placebo treatment, which will continue for 8 weeks. Subsequently participants will undergo a 4-week washout period. At the end of the washout period a second 8-week treatment block with the alternative treatment will commence.

Patients will complete a headache diary daily for at least 4 weeks prior to the baseline visit, throughout the treatment and washout periods and for 4 weeks after treatment ceases. The diary will record headache frequency, duration, intensity, pain characteristics and medication intake for comparison with baseline data.

From screening until the final study visit (over a minimum of 6 months) a total of approximately 200 mL in blood samples will be taken from each local participant.

For participants located in country or interstate locations:

The same study will be undertaken, but instead of attending the Pain and Anaesthesia Research Clinic (PARC), within the Royal Adelaide Hospital (RAH) for screening and study visits, these will be managed remotely through:

basic input from the participant's GP during the screening period correspondence with the PI and study staff via registered post, phone or Skype scheduled visits to the nearest pathology collection centre for blood biochemistry and haematology analysis

Interstate or country participants will also be exempt from collection of blood samples for biomarker analysis, hence a total of approximately 120 mL of blood samples will be taken from each interstate or country participant.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged between 18 to 65 years Migraine with or without aura, as diagnosed according to the second edition International Classification of Headache Disorders (ICHD-II) Onset of migraine before 50 years of age Headache on 15 or more days per month Migraine-like headache on 8 or more days per month, as per the IHS guidelines

Exclusion Criteria:

* Change in type or dose of migraine prophylactic medication in last 3 months
* Medication overuse headache as diagnosed according to the ICHD-IIR
* Post-traumatic headache as diagnosed according to the ICHD-II
* Other dominant chronic pain condition
* Known active inflammatory diseases such as rheumatoid arthritis
* History of recent cerebrovascular disorder
* Unable to provide written informed consent
* Unable to read and write in English
* Severe psychological/psychiatric disorders
* Recent history of significant trauma, as determined by the Principal Investigator including major surgery within the previous 2 months or major surgery planned during the treatment period
* Recent history of drug or alcohol abuse
* Any clinically significant findings on screening blood sample results
* Current malignancy
* Known hypersensitivity to ibudilast or excipients in Ketas® formulation
* Renal or hepatic impairment, defined as baseline GFR (as calculated by the Cockcroft-Gault equation) of <60 mL/min, LFTs (excluding bilirubin) > 3 times the upper limit of normal or bilirubin > 2 times the upper limit of normal
* For females of childbearing potential:

  * Pregnancy
  * Lack of adequate contraception (abstinence, double barrier method, intrauterine device, surgical sterilization (self or partner), hormonal contraceptive methods (oral, injected, or implanted)
  * Breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Primary efficacy end point | 8 weeks
  As suggested by the IHS guidelines for clinical trials in chronic migraine, the primary efficacy endpoint will be number of headache days per month with moderate or severe intensity. Study outcomes will be assessed at baseline and at weeks 2, 4 and 8 of each treatment period.
  To monitor treatment with ibudilast, blood biochemistry (including assessment of renal and hepatic including GGT function) and haematology will be assessed at baseline, and at weeks 2, 4 and 8 of each treatment period. Patients will also be screened for adverse effects via questionnaire at each visit during treatment.

SECONDARY OUTCOMES:
Secondary efficacy end points | 8 weeks
  The secondary end points assessed will include:
  * Migraine frequency (number of days with migraine of any severity/month)
  * Migraine episode frequency (number of migraine episodes/month)
  * Medication frequency (number of days acute headache medication taken/month)
  * Headache related impact on quality of life as assessed using the HIT-6
  * Cutaneous allodynia as assessed using the ASC-12
  * Biomarker levels
Serum biomarker levels | 8 weeks
  To determine if serum levels of the following potential biomarkers are able to differentiate response to treatment with ibudilast: glutamate, calcitonin gene-related peptide, glial fibrillary acidic protein and S100 calcium binding protein β.

OTHER OUTCOMES:
safety and tolerability of ibudilast | 8 weeks
  Ibudilast 40 mg or placebo twice daily for 8 weeks is effective and safe in a chronic migraine population.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Rolan, MBBS FRACP FFPM MD, Principal Investigator — School of Medical sciences, University of Adelaide, Adelaide, Australia; Parisa Gazerani, PharmD, PhD, Principal Investigator — Aalborg University
Locations (1):
- School of Medical sciences, University of Adelaide, Adelaide, Australia